CLINICAL TRIAL: NCT00841880
Title: A Prospective, Open Label, Randomized, Comparative Study of Ramipril 5mg Plus Felodipine 5mg Combined Regimen and Ramipril 10mg in Uncontrolled Hypertensive Patients
Brief Title: China Medical University Hospital (CMUH) Triapin Listing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAMFE_L_03420
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Ramipril; Felodipine

ARMS (2):
- 1 (Experimental): 2 weeks run-in of Ramipril 5 mg followed by 8 weeks of Ramipril + Felodipine
  Interventions: Drug: Ramipril + Felodipine; Drug: Ramipril
- 2 (Active Comparator): 2 weeks run-in of Ramipril 5 mg followed by 8 weeks of Ramipril 10 mg
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Ramipril + Felodipine — Ramipril 5mg + Felodipine 5mg once a day
  Arms: 1
Drug: Ramipril — 10 mg once a day
  Arms: 2
Drug: Ramipril — 5mg once a day

SUMMARY:
The objective of this study is to compare the reduction in office seated systolic blood pressure (BP) following a 8 weeks regimen of ramipril 5mg plus felodipine 5mg versus ramipril 10mg.

To compare the response rate (defined as office systolic blood pressure (SBP) / Diastolic blood pressure (DBP) reduce more than 10mmHg from baseline), and BP controlled rate (defined as SBP<140mmHg and/or DBP<90mmHg) and as SBP < 130 mmHg and /or DBP < 80 mmHg in diabetes,chronic kidney disease, known Coronary Arterial Disease (CAD) or CAD equivalent, or 10-year Framingham risk score > 10%.

To ascertain the safety and tolerability of ramipril/felodipine versus ramipril in Taiwanese population.

To compare compliance with fixed dose combination of ramipril/felodipine versus ramipril treatment.

ELIGIBILITY:
Inclusion criteria:

* Uncontrolled essential hypertension defined by office SBP/DBP > 140/90 or > 130/80 mmHg for compelling indications (diabetes mellitus, chronic kidney disease, known CAD or CAD equivalent or 10-year Framingham risk score > 10%)
* Previously untreated, or previously treated with a single antihypertensive therapy at usual dose during the last 4 weeks

Exclusion criteria:

* Female who are pregnant or breast feeding
* Office DBP> 110mmHg or office SBP >180mmHg
* Hypersensitivity to ramipril, felodipine or to any of the excipients
* Bilateral stenosis of the renal arteries, or unilateral stenosis in the single kidney
* History of intolerance to any ACE inhibitor
* History of significant renal diseases including: serum creatinine >3.0 mg/dl, or creatinine clearance <30 ml/min
* History of hereditary and/or idiopathic angioedema; or angioedema associated with previous ACEI
* Significant cardiovascular diseases, multiple drug allergies, bronchospastic disease or other malignancies requiring current medication
* Hepatic disease as indicated by any of the following: Serum Glutamooxaloacetate Transferase (SGOT) or Serum Glutamopyruvate Transferase (SGPT)>3 x upper limit of normal, or serum bilirubin > 2 x upper limit of normal
* Any other condition or therapy that, in the investigator's opinion, or as indicated in the product(s) label may pose a risk to the patient or interfere with the study objective.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Seated SBP at office | After 8-week treatment

SECONDARY OUTCOMES:
Seated DBP at office | After 4 and 8-week treatment
Seated SBP at office | After 4-week treatment
Response rate | After 4 and 8-week treatment
BP controlled rate | After 4 and 8-week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fern Lim, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Taipei, Taiwan